CLINICAL TRIAL: NCT02013895
Title: Accuracy and Reliability of GSA for Remnant Liver Function in Scheduled Hepatectomized Patients
Brief Title: Accuracy and Reliability of GSA for Remnant Liver Function
Acronym: GSA
Status: Available | Type: Expanded Access
Sponsor: Kochi University (Other)
Responsible Party: Principal Investigator, Takehiro Okabayashi, Department of Gastroenterological Surgery, Kochi University
Other Study IDs: GSA-KHSC; GSA study (Other Grant/Funding Number: Kochi Organization for Medical Reformation and Renewal)
Record Dates: First submitted 2013-12-09; First posted 2013-12-17 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-12

CONDITIONS: Both Benign and Malignant Liver Mass
Keywords: liver; surgery; liver function; GSA; ICG

INTERVENTIONS:
Device: 99mTc-GSA

SUMMARY:
Preoperative evaluation of future remnant liver function is critical for patients undergoing hepatic surgery. Overestimation of the remnant liver function can lead to life-threatening postoperative hepatic failure, and its underestimation can lead to a lost opportunity for potentially curative surgery. Conventionally, post-hepatectomy remnant liver function has been estimated preoperatively using computed tomography (CT) volumetry. CT can provide precise anatomical information, and the remnant liver volume, measured by CT volumetry, has been reported to be an effective predictor of hepatic dysfunction after hepatectomy. However, the indirect estimation of liver function by CT volumetry is reliable only when the function is assumed to be homogenous over the whole liver.

DETAILED DESCRIPTION:
99mTc-galactosyl human serum albumin (99mTc-GSA) single-photon emission CT (SPECT) was developed to facilitate investigations of regional hepatic function. A disadvantage of conventional 99mTc-GSA SPECT was poor anatomical resolution, and this newly developed SPECT has a tremendously improved anatomical resolution owing to the fusion of CT and 99mTc-GSA SPECT. Recent reports have indicated that accurate regional function, based on precise anatomical information, could be evaluated using this technique.

ELIGIBILITY:
Inclusion Criteria:

* All eligible patients were those surgically treated for hepato-biliary diseases.

Exclusion Criteria:

* Patient exclusion criteria included a body weight loss greater than 10% during the six months prior to surgery, the presence of distant metastases, or seriously impaired function of vital organs due to respiratory, renal or heart disease.

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Yasuo Shima, MD PhD, Study Chair — Kochi Health Sciences Center
Locations (1):
- Kochi Health Sciences Center, Kochi, Kochi, Japan

REFERENCES:
- [Derived] Okabayashi T, Shima Y, Morita S, Shimada Y, Sumiyoshi T, Sui K, Iwata J, Iiyama T. Liver Function Assessment Using Technetium 99m-Galactosyl Single-Photon Emission Computed Tomography/CT Fusion Imaging: A Prospective Trial. J Am Coll Surg. 2017 Dec;225(6):789-797. doi: 10.1016/j.jamcollsurg.2017.08.021. Epub 2017 Sep 11. PMID 28912030